CLINICAL TRIAL: NCT07101497
Title: Phase 2 Trial of Menin Inhibitor BN104 as Post Hematopoietic Stem Cell Transplantation Maintenance in Patients With Acute Leukemia
Brief Title: Phase 2 Trial of BN104 as Post-HSCT Maintenance in Acute Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN104 maintenance post-HSCT
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Menin Inhibitors; Post Hematopoietic Stem Cell Transplantation; Maintenance Therapy; Acute Leukemia; KMT2A Rearrangement; NPM1 Mutation; NUP98 Gene Rearrangement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BN104 maitenenace (Experimental): Eligible patients will take BN104 start from 200 or 300mg, to a targent dose of 400mg, twice daily orally, 28 days for a cycle. When used in combination with posaconazoles and voriconazole, the dose of BN104 should be reduced by 50%. A total of 24 to 36 cycles of BN104 was planned.
  Interventions: Drug: BN104 monotherapy

INTERVENTIONS:
Drug: BN104 monotherapy — BN104 will be started at 200 mg or 300mg, to a target dose of 400mg, twice daily, orally, 28 days a cycle, for a total of 24 to 36 cycles . When used in combination with posaconazoles and voriconazole, the dose of BN104 should be reduced by 50%.

SUMMARY:
This is a phase 2, open label, single arm trial. This study aims to assess the efficacy and safety of menin inhibitor BN104 as maintenance therapy in patients with acute leukemia harboring specific genetic alterations who have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Eligible patients will be screened at 30-180 days post allo-HSCT. Participants will take BN104 100-200mg orally, twice a day, 28 days a cycle for 24-36 cycles. The primary endpoint is 2-year relapse-free survival rate since enrollment. The secondary endpoints included overall survival, event-free survival, cumulative incidence of relapse, non relpase related mortality and safety.

DETAILED DESCRIPTION:
AML with KMT2A rearrangements are grouped as a high risk subtype. Allogenic hematopoietic stem cell transplantation is the only curative strategy for this subtype. However, patients with KMT2A rearrangements have a high incidence of relapse rates. BN104 is a menin inhibitor. It has shown promising remission rates in patients with relpased or refractory patients haboring specific fusions including KMT2A rearrangements. The role of BN104 in post-HSCT maintenance therapy remains unknown.

This is a phase 2, open label, single arm trial. This study aims to assess the efficacy and safety of menin inhibitor BN104 as maintenance therapy in patients with acute leukemia harboring specific genetic alterations who have undergone allogeneic hematopoietic stem cell transplantation (allo-HSCT).

Eligible patients will be screened at 30-180 days post allo-HSCT. Participants will take BN104 100-200mg orally, twice a day, 28 days a cycle for 24-36 cycles. The primary endpoint is 2-year relapse-free survival rate since enrollment. The secondary endpoints included overall survival, event-free survival, cumulative incidence of relapse, non relpase related mortality, incidence of acute and chronic graft versus host diseas, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* Adult and adolescent patients aged ≥12 years who must weight ≥35 kg.
* Diagnosed with acute myeloid leuekmia, acute lymphoblastic leukemia or ambiguous acute leukemia according to the World Health Organization classification of hematologic neoplams (WHO 2022).
* Intermediate or high risk accroding to the ELN risk stratification.
* Harboring one of the following genetic aberrations: a. somatic NPM1 mutation (without FLT3-ITD/TKD co-mutations); b. KMT2A rearrangement/KMT2A-PTD; c. NUP98 rearrangement; d. other genetic alterations dependent on menin-KMT2A.
* Received allogenic hematopoietic stem cell transplantation within 30-180 days at the initiation of BN104 maintenance therapy.
* Achieved full donor chimerism and hematologic recovery, with acute neuthrophil count (ANC) ≥1.0×10⁹/L, platelets ≥75×10⁹/L (no red blood cells /platelets transfusion within 7 days, no G-CSF or GM-CSF within 72 hours).
* Complete hematological remission (CHR) after first allo-SCT. CHR must be confirmed by bone marrow analysis within 14 days before entering the study (CHR criteria are: "< 5% marrow blasts, no peripheral blasts, blood platelet count > 75×10⁹/L, WBC count > 3.5 G/L, ANC ≥ 1.0×10⁹/L).
* No extramedullary leukemia.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-2.
* Adequate organ function
* Provided informed consent by all patients and the guardians ( aged 12-17 years).
* Written informed consent.
* ECOG ≥ 2.

Exclusion Criteria:

* Complicated with active and uncontrolled infections.
* Activation of virus, (e.g., CMV viremia with CMV DNA copies > 400 copies/ml, EBV viremia with EBV DNA copies > 400 copies/ml, and proof of activation of adenovirus and Human Parvovirus B19 ).
* Activation of hepatitis B, hepatitis C, or human immunodeficiency virus.
* Cardiac disease as followings: a. inherited long QT syndrome. b. Congestive heart failure with NYHA ≥ grade 2.
* ≥ grade 2 acute GVHD or ≥ grade 3 chronic GVHD which requiring systemic therapy.
* Have received other maintenance therapies (e.g., hypomethylating agents, targetd drugs such as Bcl-2 inhibitors, FLT3 inhibitors, IDH1/2 inhibitors, interferon, interleukin-2, donor lymphocyte infusion and chemotherapy).
* History of other malignancies which needed systemic treatment (excluding those in stable remission without maintenance therapy).
* Any gastrointestinal condition that may interfere with oral drug intake or absorption (e.g., dysphagia, gastroparesis, uncontrolled chronic diarrhea, intestinal graft versus host disease.
* Pregnancy, breastfeeding
* Hypersensitivity to BN104.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year rate of RFS | 2 years
  It is measured as the proportions of numbers of patients with hematologic relapse to the numbers of the overall enrolled patients at 2 years from the first day of taking BN104 post allo-HSCT.

SECONDARY OUTCOMES:
OS | 2 years
  Overall survival (OS): It is measured from the date of the first day of taking BN104 post allo-HSCT to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
EFS | 2 years
  Event-freesurvival: It is measured from he date from the first day of taking BN104 post allo-HSCT to the first documented hematologic relapse, initiation of other maintenance therapy stragies such as hypomethylation agents, interferon, donor lymphocyte infusion, Bcl-2 inhibitor or death from any cause. Patients who die without evidence of relapse are typically censored at the last disease-free assessment.
CIR | 2 years
  Cumulative incidence of relapse (CIR): It is measured as the estimated rate of hematologic relapse or extramedullary relapse since the first day of taking BN104 post allo-HSCT.
NRM | 2 years
  non-relapse mortality (NRM): It is measured the probability of death attributable to treatment-related complications or comorbidities, excluding disease relapse/progression since the first day of taking BN104 post allo-HSCT.
Incidence and severity of GVHD | 2 years
  Incidence and severity of acute and chronic GVHD since the first day or taking BN104 post allo-HSCT.

OTHER OUTCOMES:
Pre-/post-transplant MRD dynamics | 2 years
  Serial monitoring results of measurable residual disease status detected by qPCR or Ig/TR rearrangements since the first day of taking BN104
Impact of BN104 on immune recovery | 2 years
  Serial monitoring results of Immunoglobulin levels, T-cell subsets or cytokine profiling since the first day of taking BN104 post allo-HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Su-ning Chen, M.D., Principal Investigator — (0086)13814881746
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China